CLINICAL TRIAL: NCT00481949
Title: What is the Physiologic and Clinical Relevance of Oesophagogastric Junction Distensibility? Studies Using Endo-Flip and 96 Hour Wireless pH System
Brief Title: Assessment of Gastro-esophageal Reflux Using Endo-Flip vs Bravo
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Mark Fox, GuysThomasNHS
Other Study IDs: 05/20702/84
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Heartburn; Gastro-esophageal Reflux
Keywords: Gastro-oesophageal reflux disease; pH measurement; symptom association; wireless pH monitoring system; Functional Heartburn; Gastro-esophageal reflux disease
MeSH Terms: conditions — Heartburn; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsies taken at the gastro-oesophageal junction will be sent to histology lab and analysed as per routine histology specimens. These will be stored as all samples at our hospital are stored and only results reported by the appointed histologist will be used for analysis.
Oversight: Data Monitoring Committee: No

SUMMARY:
Monitoring oesophageal pH provides a definitive diagnosis of patients with gastro-oesophageal reflux disease (GORD), especially those in whom the association between reflux and symptoms is uncertain and those under consideration for anti-reflux surgery. Standard ambulatory investigation is normally performed by naso-oesophageal catheter however this is associated with considerable discomfort and in turn altered behaviour which reduces reflux provoking activities. Furthermore results of catheter based ambulatory pH studies are compromised by the high variability of acid exposure in patients with suspected GORD.

Prolonging pH measurements by the catheter-free Bravo™ system from 24 to 48 and 96hrs significantly improves the consistency (reliability) and reproducibility of diagnoses based on oesophageal acid exposure, as well as the ability to associate acid reflux to symptom episodes. This improves diagnosis especially in those with intermittent symptoms.

However pH monitoring does not provide a direct assessment of the underlying pathophysiology. Incompetence of the oesophago-gastric junction (OGJ) related to disruption of its structure and function is considered to be the most important cause of GORD. A more relevant assessment of the reflux barrier may be its distensibility (i.e. the ease with which the OGJ is opened to allow retrograde passage of gastric contents); however this is not assessed by current clinical investigations.

Endo-FLIP (Crospon Medical Devices) is a new tool which assesses OGJ structure and function, and appears to provide relevant information regarding its distensibility and competence.

This study applies to using Endo-Flip to record OGJ distensibility and Bravo to record acid exposure and symptom association in patients with reflux symptoms. The variability of pH measurements and symptoms and diagnostic accuracy will be assessed over 96hrs. Endo-FLIP results will then be compared against Bravo. The outcome of post investigation therapy will then be compared with Endo-Flip and Bravo results to assess if baseline testing can predict the outcome of acid suppression therapy.

Study Hypothesis

1. There is a positive, continuous association between OGJ distensibility measured by Endo-FLIP on % acid exposure assessed by prolonged Bravo pH monitoring
2. The results of Endo-FLIP and prolonged Bravo predict treatment outcome of a trial of proton pump inhibitor therapy

DETAILED DESCRIPTION:
This is a single centre study of patients (n=60) referred for investigation of reflux symptoms. Each patient is investigated by Endo-FLIP™, endoscopy, and 96 hour Bravo™ pH monitoring off acid suppressant medication.

After calibration the Endo-FLIP catheter will be inserted orally or nasally until the liquid-filled compliant bag at the distal segment of the catheter (which houses 16 impedance sensors) straddles the OGJ. Stepwise bag distensions of 10, 20 and 30 ml will then be conducted and the associated intra-bag pressure measured. The Endo-FLIP display will allow real-time imaging of OGJ intra-luminal geometry during distension. Intra-bag pressure and CSA at the impedance planimetry segment best localized within the OGJ will be reported as mean ± SEM.

An endoscopy will then be performed to confirm the position of the squamo-columnar junction (SCJ). Images will be taken of the SCJ using standard white light and narrow band imaging. Then 2 x 2 biopsies from the SCJ and 2 cm proximally will be taken. In conclusion, the Bravo® delivery system will be passed orally with the patient lying in the left lateral decubitus position and the capsule will be deployed 6 cm proximal to the SCJ after 1 minute of suction to stabilize the position.

After 2 measurements for 48 hours (separated by a battery change) the patient will return the receiver for the final download and analysis. In addition to pH measurement and symptom documentation during the 96hr period, pepsin lateral flow tests (Technostics, Hull, UK) will be performed by collecting expectorated saliva on returning to the lab on day 2 and day 4. Patients will also be provided with two further kits to be used if and when they experience symptoms during the 4 day study.

The primary outcome assessment of oesophageal acid exposure will be percent time pH<4 over the measurement period (e.g. 24, 48 or 96h). Other parameters that will be analysed are the number of reflux events and the association of these events with symptoms recorded on the Bravo™ receiver. The presence or absence of pepsin in expectorated saliva will also be assessed.

All subjects will complete a quality of life assessment (SF-36). Symptom severity will be assessed at baseline and at follow-up and will be documented by validated questionnaires (Eraflux) before and after resumption of routine acid reducing therapy. Those that undergo anti-reflux surgery will also be followed up at 3 and 6 months.

LOS distensibility measurements using Endo-FLIP will also be collected in those diagnosed with achalasia on manometry in order to be used as reference values for the Bravo study.

Patient symptoms will be reviewed at baseline off treatment and again after six weeks of returning back onto their standard acid reducing medication. Patients referred for anti-reflux surgery will be reviewed 3 and 6 months after the procedure.

This is a prospective study of 60 consecutive patients referred for the investigations typical reflux symptoms (power calculations to allow comparison of 24hr vs. 48hr pH testing).

Analysis

Bravo:

1. Retrospective analysis: Formal statistical analysis of the pH and symptom database that was collected prospectively over the last 4 years (contains >200 Bravo pH studies). This will establish the correlation between pH results from 24, 48 and 96hr monitoring with clinical variables (e.g. severity of reflux symptoms, symptom association) and outcome (e.g. response to PPI, response to fundoplication).
2. Prospective analysis: The day-to-day variability of pH measurements will be calculated. Patients will be classified by acid exposure (abnormal: >4.2% time pH<4) and symptom index (positive SI: >50% association of reflux events and any symptom) during each 24hr and 48hr test period. The reproducibility and accuracy of 24hr vs. 48hr pH testing will be assessed with 96hr results as the reference standard.

Endo-Flip: Stepwise bag distensions of 10, 20 and 30 ml will be conducted and the associated intra-bag pressure measured. The Endo-FLIP display will allow real-time imaging of OGJ intraluminal geometry during distension. The primary outcome assessment of OGJ distensibility will be the intra-bag pressure and cross-sectional area at the impedance planimetry segment best localized within the LOS as mean ± SEM for each consecutive volume distension. The correlation of OGJ distensibility with oesophageal acid exposure will then be assessed.

The correlation and interaction between OGJ distensibility, acid exposure, reflux-symptom association and symptom characteristics (e.g. severity and predominant symptom) at baseline and on treatment will be assessed by co-variant regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written, fully informed consent to undergo mechanistic procedures: Endo-FLIP, endoscopy and biopsy, 4 day wireless pH monitoring by the Bravo system
* All subjects should be off acid suppression medication (e.g. PPI, H2RA) for at least 5 days prior to endoscopy

Exclusion Criteria:

* Significant gastrointestinal symptoms or disease other than reflux
* Previous upper GI surgery or interventions such as oesophageal dilatations
* Predominant symptoms of motility disorders, e.g. dysphagia
* Presence of major oesophageal dysmotility on manometry, e.g. achalasia
* Significant co-morbidity requiring ongoing treatment or investigation
* Physical, neurological or psychiatric conditions preventing repeated visits to hospital or compliance with study procedures (e.g. physical impairment/reduced mobility)
* Pregnant at the time of enrolment
* No haematological abnormalities (no anticoagulants)
* No medications influencing gastrointestinal function within 3 days of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with typical reflux symptoms (heartburn, acid regurgitation)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic reliability of prolonged wireless pH monitoring and comparison oesophago-gastric junction distensibility | 1 year
  1. To confirm improved diagnostic reliability and accuracy of prolonged pH measurement by the Bravo™ system in a large, prospective clinical trial
  2. To confirm that there is a positive, continuous association between oesophago-gastric junction (OGJ) distensibility measured by Endo-FLIP on percentage acid exposure assessed by prolonged Bravo-pH monitoring

SECONDARY OUTCOMES:
Prediction of treatment outcome with Endo-Flip and Bravo | 2 years
  To confirm that the results of Endo-FLIP and prolonged Bravo-pH monitoring can predict treatment outcome of a trial of proton pump inhibitor therapy:
  1. Patients with high OGJ distensibility and high reflux-symptom association with acid regurgitation or cough complain of persistent regurgitation of gastric contents on treatment.
  2. Patients with low OGJ distensibility and high reflux-association with heartburn complain of persistent heartburn
  3. Patients with low OGJ distensibility and low reflux-association with any symptom complain of atypical and dyspeptic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fox, MD, Principal Investigator — Honorary Consultant and Senior Lecturer
Locations (1):
- Oesophageal Laboratory, GSTT, London, London, United Kingdom